CLINICAL TRIAL: NCT03296800
Title: A Phase 1, Open-Label, Non-Randomized, Fixed-Sequence Composite Study to Evaluate the Effects of Probenecid, Rifampin, and Verapamil on the Pharmacokinetics and Pharmacodynamics of Bexagliflozin in Healthy Subjects
Brief Title: Study to Evaluate Effects of Probenecid, Rifampin and Verapamil on Bexagliflozin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Theracos (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: THR-1442-C-454
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bexagliflozin; Probenecid; Rifampin; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Bexagliflozin/probenecid (Experimental): Sixteen healthy subjects were dosed with bexagliflozin, qd and/or probenecid tablets, 500 mg, bid, in sequential order as follows: on Day 1 subjects took bexagliflozin; on Days 3 and 4 subjects took probenecid, bid; on Day 5 subjects took one bexagliflozin, and probenecid, bid; and on Day 6 subjects took probenecid tablets, 500 mg, bid.
  Interventions: Drug: Bexagliflozin; Drug: Probenecid
- Bexagliflozin/rifampin (Experimental): Sixteen healthy subjects were dosed with bexagliflozin, qd and/or 600 mg of rifampin daily in sequential order as follows: on Day 1 subjects took one bexagliflozin tablet; on Days 3 to 5, subjects took rifampin once daily; on Day 6 subjects took one bexagliflozin tablet and rifampin; and on Day 7 subjects took rifampin.
  Interventions: Drug: Bexagliflozin; Drug: Rifampin
- Bexagliflozin/verapamil (Experimental): Sixteen healthy subjects were dosed with bexagliflozin, and/or verapamil tablets, 120 mg in sequential order as follows: on Day 1 subjects took one bexagliflozin tablet, on Day 4 subjects took one verapamil tablet, 1 hour before taking a bexagliflozin tablet.
  Interventions: Drug: Bexagliflozin; Drug: Verapamil

INTERVENTIONS:
Drug: Bexagliflozin — Bexagliflozin 20 mg, tablet; qd
  Other Names: EGT0001442, EGT0001474
Drug: Probenecid — Probenecid tablets, 500 mg; bid
  Other Names: Probalan
  Arms: Bexagliflozin/probenecid
Drug: Rifampin — Rifampin, 600 mg (2 x 300 mg capsules); qd
  Other Names: Rifadin
  Arms: Bexagliflozin/rifampin
Drug: Verapamil — Verapamil hydrochloride tablet, 120 mg; qd
  Other Names: Verelan
  Arms: Bexagliflozin/verapamil

SUMMARY:
The purpose of this study is to examine the drug-drug interaction when given the study drug, bexagliflozin, with three commonly prescribed medications, probenecid, verapamil or rifampin. The study is to evaluate how safe the study drug is and how well the study drug is tolerated when taken with probenecid, verapamil or rifampin.

DETAILED DESCRIPTION:
In this study, a total of 48 healthy subjects were enrolled and assigned to one of three groups of 16 subjects. Each group participated in an open-label, non-randomized, fixed-sequence studies to assess potential interaction of bexagliflozin tablets, 20 mg with probenecid, rifampin or verapamil.

Sequence 1: Bexagliflozin/probenecid Sixteen healthy subjects were dosed with bexagliflozin, qd and/or probenecid tablets, 500 mg, bid, in sequential order as follows: on Day 1 subjects took bexagliflozin; on Days 3 and 4 subjects took probenecid, bid; on Day 5 subjects took one bexagliflozin, and probenecid, bid; and on Day 6 subjects took probenecid tablets, 500 mg, bid.

Sequence 2: Bexagliflozin/rifampin Sixteen healthy subjects were dosed with bexagliflozin, qd and/or 600 mg of rifampin daily in sequential order as follows: on Day 1 subjects took one bexagliflozin tablet; on Days 3 to 5, subjects took rifampin once daily; on Day 6 subjects took one bexagliflozin tablet and rifampin; and on Day 7 subjects took rifampin.

Sequence 3: Bexagliflozin/verapamil Sixteen healthy subjects were dosed with bexagliflozin, and/or verapamil tablets, 120 mg in sequential order as follows: on Day 1 subjects took one bexagliflozin tablet, on Day 4 subjects took one verapamil tablet, 1 hour before taking a bexagliflozin tablet.

ELIGIBILITY:
Subjects meeting the following Criteria were included::

1. Between 18 and 55 years of age at screening, inclusive, and in good health based on medical history, physical examination, electrocardiogram and routine laboratory tests.
2. Had a body-mass index (BMI) between 18.0 kg/m2 and 32.0 kg/m2 at screening, inclusive.
3. Abstained from tobacco consumption for at least 3 months prior to screening.
4. Had adequate venous access at multiple sites in both arms.
5. Willing and able to be confined to the clinical research facility as required by the protocol.
6. Able to comprehend the explanation of the informed consent and willing to provide written informed consent in accordance with institutional and regulatory guidelines.

Subjects who met any of the following criteria were excluded from the study:

1. A clinically significant history of allergy to drugs or latex (at the Investigator's discretion.)
2. A history of alcohol or drug dependence in the last 12 months.
3. A history of donation of 400 mL of whole blood within two months, 200 mL of whole blood within one month, or blood components within 14 days prior to the first dose.
4. A history of prescription or over-the-counter (OTC) drug use within 14 days prior to the first dose.
5. A history of vitamin preparation or supplement use (including St. John's Wort and ginseng) within 14 days prior to the first dose.
6. A history of strenuous physical activity within 72 hours prior to dosing.
7. A history of exposure to an investigational drug within 30 days or 7 half-lives of the investigational drug, whichever was longer, prior to the first dose of investigational drug in this trial.
8. A history of prior exposure to EGT0001474 or bexagliflozin at any time, or of exposure to any other SGLT2 inhibitors within 3 months from screening or of participation in previous bexagliflozin clinical trials.
9. A history of consumption of probenecid, rifampin, or verapamil within 3 months of screening.
10. A screening ECG that demonstrated any one of the following: heart rate >100 bpm, QRS >120 msec, QTc >470 msec (corrected by Bazett's formula), PR >220 msec (a subject with PR >220 msec was generally to be excluded, but exceptions may have been allowed at the discretion of the Investigator), or any clinically significant arrhythmia.
11. A sitting blood pressure that was above 140/90 mmHg at screening. If the sitting blood pressure at screening was above 140/90 mmHg, one repeat measurement could have been taken. Subjects were to be excluded if the repeated sitting blood pressure was above 140/90 mmHg, but exceptions may have been allowed at the discretion of the Investigator.
12. A positive result for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or for urinary drug or cotinine tests.
13. A history of human immunodeficiency virus (HIV) infection.
14. A history of febrile illness within 5 days prior to the first dose of investigational drug.
15. A history of vaccination (with the exception of the flu vaccine) within 30 days prior to the first dose of investigational drug.
16. An estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m2 or a history of kidney transplant.
17. If male, who was not surgically sterile, unwilling to refrain from donating sperm, and/or unwilling to use appropriate birth control when engaging in sexual intercourse for a period of 30 days after discharge from the clinic.
18. Female subjects who were surgically sterile (i.e., have undergone partial or full hysterectomy, or bilateral oophorectomy) or postmenopausal were eligible if they tested negative on a urine pregnancy test.
19. Evidence of anemia if selected for probenecid study.
20. Evidence of abnormal liver function tests (total bilirubin >1.5 x upper limit of normal [ULN]); or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2.5 x ULN.
21. If selected for the rifampin study, unwilling to refrain from the use of soft contact lenses during the study.
22. Unwilling to forgo consumption of alcohol 72 hours pre admission and throughout the study.
23. Unwilling to forgo consumption of grapefruit and grapefruit products from 7 days prior to dosing through discharge from the clinic.
24. A history of recurrent yeast or urinary tract infections or any such infections in the 6 months prior to first dose.
25. A history of gout, glucose-6-phosphate dehydrogenase deficiency, or nephrolithiasis if a candidate for the probenecid study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-09-27 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mason Freeman, M.D., Study Director — Massachusetts General Hospital
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Bexagliflozin, Then Probenecid, Then Bexagliflozin and Probenecid: Subjects were dosed with bexagliflozin tablets, 20 mg, qd and/or probenecid tablets, 500 mg, bid, in sequential order as follows: on Day 1 subjects took bexagliflozin; on Days 3 and 4 subjects took probenecid, bid; on Day 5 subjects took one bexagliflozin, and probenecid, bid; and on Day 6 subjects took probenecid tablets, 500 mg, bid.
- Bexagliflozin, Then Rifampin, Then Bexagliflozin and Refampin: Subjects were dosed with bexagliflozin tablets, 20 mg, qd and/or 600 mg of rifampin daily in sequential order as follows: on Day 1 subjects took one bexagliflozin tablet; on Days 3 to 5, subjects took rifampin once daily; on Day 6 subjects took one bexagliflozin tablet and rifampin; and on Day 7 subjects took rifampin.
- Bexagliflozin, Then Verapamil and Bexagliflozin: Subjects were dosed with bexagliflozin tablets, 20 mg, and/or verapamil tablets, 120 mg in sequential order as follows: on Day 1 subjects took one bexagliflozin tablet, on Day 4 subjects took one verapamil tablet, 1 hour before taking a bexagliflozin tablet.
Period: Overall Study
Arm/Group | Bexagliflozin, Then Probenecid, Then Bexagliflozin and Probenecid | Bexagliflozin, Then Rifampin, Then Bexagliflozin and Refampin | Bexagliflozin, Then Verapamil and Bexagliflozin
Started | 16 | 16 | 16
Completed | 16 | 16 | 16
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bexagliflozin, Then Probenecid, Then Bexagliflozin and Probenecid: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Probenecid: Probenecid tablets, 500 mg; bid
- Bexagliflozin, Then Rifampin, Then Bexagliflozin and Refampin: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Rifampin: Rifampin 600 mg (2 x 300 mg capsules); qd
- Bexagliflozin, Then Verapamil and Bexagliflozin: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Verapamil: Verapamil hydrochloride tablets, 120 mg; qd
- Total: Total of all reporting groups
Arm/Group | Bexagliflozin, Then Probenecid, Then Bexagliflozin and Probenecid | Bexagliflozin, Then Rifampin, Then Bexagliflozin and Refampin | Bexagliflozin, Then Verapamil and Bexagliflozin | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (9.69) | 35.3 (10.72) | 37.8 (11.24) | 37.2 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 12
  Male | 13 | 11 | 12 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 8 | 26
  Not Hispanic or Latino | 6 | 8 | 8 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 5 | 12
  White | 11 | 14 | 11 | 36
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 81.3 (10.59) | 74.1 (11.31) | 78.9 (9.21) | 78.7 (10.57)
Height [Mean (Standard Deviation); unit: cm] | 170.9 (8.28) | 169.2 (8.38) | 172.1 (10.17) | 170.7 (8.88)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.8 (2.73) | 25.9 (3.31) | 26.7 (2.46) | 27.0 (3.50)

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Plasma Concentration)
Description: Whole venous blood samples of 3 mL were collected from a peripheral vein prior to dosing and at 1, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 36, and 48 h after administration of bexagliflozin; On Day 1 and Day 5 for Study 1, Day 1 and Day 6 for Study 2, Day 1 and Day 4 for Study 3. The pharmacokinetic parameters were estimated from the bexagliflozin plasma concentration data for each subject by non-compartmental analysis (NCA).
Time Frame: Up to 48 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Study 1: Bexagliflozin Alone; Study 2: Bexagliflozin Alone; Study 3: Bexagliflozin Alone: Bexagliflozin tablets, 20 mg; qd
- Study 1: Bexagliflozin and Probenecid: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Probenecid: Probenecid tablets, 500 mg; bid
- Study 2: Bexagliflozin and Rifampin: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Rifampin: Rifampin 600 mg (2 x 300 mg capsules); qd
- Study 3: Bexagliflozin and Verapamil: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Verapamil: Verapamil hydrochloride tablets, 120 mg; qd
Arm/Group | Study 1: Bexagliflozin Alone | Study 1: Bexagliflozin and Probenecid | Study 2: Bexagliflozin Alone | Study 2: Bexagliflozin and Rifampin | Study 3: Bexagliflozin Alone | Study 3: Bexagliflozin and Verapamil
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
ng/mL | 161.675 (28.673) | 193.366 (22.098) | 97.811 (53.903) | 117.001 (60.097) | 159.355 (35.396) | 169.000 (24.727)
Statistical Analysis 1: Comparison: Study 1: Bexagliflozin Alone vs Study 1: Bexagliflozin and Probenecid; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Point Estimate (%) = 118.66, 90% CI 2-sided [111.12 to 126.72] — Point Estimate is the estimated ratio of exponentiated mean difference of log-transformed PK parameter from ANOVA. Confidence interval is obtained from ANOVA with treatment as a fixed effect, and subject as a random effect
Statistical Analysis 2: Comparison: Study 2: Bexagliflozin Alone vs Study 2: Bexagliflozin and Rifampin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Point Estimate (%) = 119.62, 90% CI 2-sided [94.39 to 151.59]; Point Estimate is the estimated ratio of exponentiated mean difference of log-transformed PK parameter from ANOVA. Confidence interval is obtained from ANOVA with treatment as a fixed effect, and subject as a random effect
Statistical Analysis 3: Comparison: Study 3: Bexagliflozin Alone vs Study 3: Bexagliflozin and Verapamil; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Point Estimate (%) = 106.05, 90% CI 2-sided [88.81 to 126.65]; [other analysis details as in outcome 1, analysis 2]

2. Primary Outcome: Tmax (Time of Maximum Observed Plasma Concentration)
Description: as for outcome 1
Time Frame: Up to 48 hours
Measure: Median (Full Range); unit: hours
Groups:
- Bexagliflozin/Probenecid: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Probenecid: Probenecid tablets, 500 mg; bid
- Bexagliflozin/Rifampin: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Rifampin: Rifampin 600 mg (2 x 300 mg capsules); qd
- Bexagliflozin/Verapamil: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Verapamil: Verapamil hydrochloride tablets, 120 mg; qd
Arm/Group | Bexagliflozin/Probenecid | Bexagliflozin/Rifampin | Bexagliflozin/Verapamil
Number analyzed (Participants) | 16 | 16 | 16
hours
  Bexagliflozin alone | 2.000 [2.000 to 4.000] | 2.000 [2.000 to 4.083] | 3.0 [2.000 to 8.000]
  Bexagliflozin + additional drug | 3.000 [2.000 to 4.017] | 2.000 [1.017 to 4.000] | 3.000 [2.000 to 4.000]

3. Primary Outcome: T1/2 (Apparent Terminal Elimination Half-life)
Description: as for outcome 1
Time Frame: Up to 48 hours
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Bexagliflozin/Probenecid | Bexagliflozin/Rifampin | Bexagliflozin/Verapamil
Number analyzed (Participants) | 16 | 16 | 16
hours
  Bexagliflozin alone | 12.090 (35.950) | 12.190 (36.966) | 10.709 (44.103)
  Bexagliflozin + additional drug | 13.894 (24.806) | 5.318 (49.740) | 11.675 (48.222)

4. Primary Outcome: AUC0-inf (Area Under the Plasma Concentration-time Curve From Time 0 to Infinity)
Description: as for outcome 1
Time Frame: Up to 48 hours
Population: AUC0-t (from time 0 to time T) was used instead of AUC0-inf for Study 2 since AUC0-inf was not reported
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Groups:
- Study 1: Bexagliflozin/Probenecid: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Probenecid: Probenecid tablets, 500 mg; bid
- Study 2: Bexagliflozin/Rifampin: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Rifampin: Rifampin 600 mg (2 x 300 mg capsules); qd
- Study 3: Bexagliflozin/Verapamil: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Verapamil: Verapamil hydrochloride tablets, 120 mg; qd
Arm/Group | Study 1: Bexagliflozin Alone | Study 1: Bexagliflozin/Probenecid | Study 2: Bexagliflozin Alone | Study 2: Bexagliflozin/Rifampin | Study 3: Bexagliflozin Alone | Study 3: Bexagliflozin/Verapamil
Number analyzed (Participants) | 15 | 16 | 16 | 16 | 16 | 16
hr*ng/mL | 1118.741 (23.290) | 1583.188 (23.676) | 698.254 (43.945) | 601.334 (49.870) | 1025.101 (25.746) | 1003.931 (21.571)
Statistical Analysis 1: Comparison: Study 1: Bexagliflozin Alone vs Study 1: Bexagliflozin/Probenecid; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Point Estimate (%) = 140.98, 90% CI 2-sided [131.39 to 151.26] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Study 2: Bexagliflozin Alone vs Study 2: Bexagliflozin/Rifampin; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Point Estimate (%) = 86.12, 90% CI 2-sided [70.24 to 105.59] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Study 3: Bexagliflozin Alone vs Study 3: Bexagliflozin/Verapamil; Geometric LS Mean was used as PK parameters; Test type: Equivalence — The acceptance range for bioequivalence is 80.0 - 125.00%; Point Estimate (%) = 97.93, 90% CI 2-sided [90.26 to 106.26] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Urinary Glucose Excretion 0-48 hr
Description: Pre-dose urine samples were collected from -12 to 0 h for baseline measurement of pharmacodynamic parameters. Post-dose urine samples were collected without preservative in four batches: 0 to 12 h, 12 to 24 h, 24 to 36h, and 36 to 48 h after dosing. Urine aliquots were prepared from well mixed collections for the assessment of pharmacodynamics.
Time Frame: 0 to 48 hours
Population: Only subjects with data in the specific category is included
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Study 1: Bexagliflozin Alone | Bexagliflozin/Probenecid | Study 2: Bexagliflozin Alone | Bexagliflozin/Rifampin | Study 3: Bexagliflozin Alone | Bexagliflozin/Verapamil
Number analyzed (Participants) | 16 | 16 | 16 | 16 | 16 | 16
g
  Pre-dose (-12 - 0 hours) | 0.02 (0.024) | 0.47 (1.160) | 0.02 (0.014) | 0.12 (0.180) | 0.02 (0.018) | 1.37 (1.476)
  0 - 12 hours post-dose: number analyzed (Participants) | 15 | 16 | 16 | 16 | 16 | 16
  0 - 12 hours post-dose | 25.04 (5.579) | 25.90 (5.214) | 31.50 (9.272) | 31.40 (7.363) | 31.14 (5.814) | 31.46 (14.835)
  12 - 24 hours post-dose | 21.28 (7.347) | 20.92 (4.358) | 19.43 (6.863) | 15.72 (7.259) | 22.30 (3.933) | 20.51 (5.940)
  24 - 36 hours post-dose: number analyzed (Participants) | 15 | 16 | 16 | 16 | 16 | 16
  24 - 36 hours post-dose | 22.04 (7.136) | 22.10 (6.826) | 21.51 (7.668) | 16.32 (6.370) | 24.54 (6.517) | 20.94 (6.745)
  36 - 48 hours post-dose | 11.15 (5.447) | 9.53 (3.114) | 6.99 (3.440) | 3.41 (2.318) | 11.31 (4.997) | 4.78 (2.941)
  0 - 24 hours post-dose: number analyzed (Participants) | 15 | 16 | 16 | 16 | 16 | 16
  0 - 24 hours post-dose | 47.73 (9.125) | 46.82 (8.530) | 50.93 (15.606) | 47.12 (13.790) | 53.44 (8.712) | 51.97 (13.658)
  0 - 48 hours post-dose: number analyzed (Participants) | 15 | 16 | 16 | 16 | 16 | 16
  0 - 48 hours post-dose | 81.67 (16.083) | 78.44 (15.653) | 79.43 (24.490) | 66.86 (19.564) | 89.29 (16.461) | 77.69 (16.497)

ADVERSE EVENTS:
Time Frame: The adverse event data were collected from Day 0 up to Day 7 for study 1, Day 0 up to Day 8 for study 2 and Day 0 up to Day 6 for study 3 after drug administration
Groups:
- Study 1: Bexagliflozin Alone; Study 2: Bexagliflozin Alone; Study 3: Bexagliflozin Alone: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
- Study 2: Bexagliflozin and Rrifampin: Bexagliflozin: Bexagliflozin tablets, 20 mg; qd
  Rifampin: Rifampin 600 mg (2 x 300 mg capsules); qd
Arm/Group | Study 1: Bexagliflozin Alone | Study 1: Bexagliflozin and Probenecid | Study 2: Bexagliflozin Alone | Study 2: Bexagliflozin and Rrifampin | Study 3: Bexagliflozin Alone | Study 3: Bexagliflozin and Verapamil
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 1/16 | 0/16 | 0/16 | 2/16 | 0/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study 1: Bexagliflozin Alone (N=16) | Study 1: Bexagliflozin and Probenecid (N=16) | Study 2: Bexagliflozin Alone (N=16) | Study 2: Bexagliflozin and Rrifampin (N=16) | Study 3: Bexagliflozin Alone (N=16) | Study 3: Bexagliflozin and Verapamil (N=16)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal sounds abnormal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator has no right to publish the trial results.

DOCUMENTS (2):
  • Study Protocol (2017-08-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT03296800/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03296800/SAP_001.pdf